CLINICAL TRIAL: NCT06736431
Title: Bringing Advocacy Via Digital Guide to the Emergency Department (Project BADGE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sara Heinert, PhD, MPH, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2024001476
Record Dates: First submitted 2024-12-13; First posted 2024-12-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Text-based platform (Experimental): Text-based resource referral platform with diabetes educational materials
  Interventions: Behavioral: Text-based resource referral platform with diabetes educational materials

INTERVENTIONS:
Behavioral: Text-based resource referral platform with diabetes educational materials — Text-based resource referral platform with diabetes educational materials

SUMMARY:
The pilot study of Project BADGE will focus on emergency department (ED) patients with diabetes, which has significant disparities in prevalence and mortality for underserved populations. The objective is to determine the effect of a text-based resource referral platform with diabetes educational materials on patient diabetes knowledge, diabetes distress, diabetes self-care activities, and acceptability and feasibility of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (18+) ED/observation unit patients
2. Have poorly controlled or new onset diabetes (hyperglycemia or Diabetic ketoacidosis (DKA))
3. Speak English or Spanish
4. Has a cell phone able to send and receive text messages

Exclusion Criteria:

1) Intubated patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress | Baseline, 3 months
  2-item Diabetes Distress Scale (DDS2)- if positive on DDS2, will complete DDS17 (On a scale of 1- "not a problem" to 6- "a very serious problem.")
Diabetes Knowledge | Baseline, 3 months
  Diabetes Knowledge Questionnaire, with response choices of Yes, No, or I Don't Know
Diabetes Self-Care | Baseline, 3 months
  Diabetes Self-Care Assessment, which asks about ask you about diabetes self-care activities during the past 7 days.
Doctor Visit | 3 months
  Did the patient attend a doctor appointment?

SECONDARY OUTCOMES:
Intervention Acceptability | 3 months
  Acceptability of Intervention Measure (AIM) on a scale of 1 (completely disagree) to 5 (completely agree)
Intervention Feasibility | 3 months
  Feasibility of Intervention Measure (FIM) on a scale of 1 (completely disagree) to 5 (completely agree)

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided